CLINICAL TRIAL: NCT05861700
Title: The Effect of Bicarbonate Profiling in Dialysis Fluid on Phosphate Removal During Hemodialysis and Blood pH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Collaborators: University of Warsaw (Other); Polish Academy of Sciences (Other)
Responsible Party: Principal Investigator, Monika Wieliczko, Clinical Doctor, Medical University of Warsaw
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KB/91/2018
Record Dates: First submitted 2023-05-06; First posted 2023-05-17 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Phosphorus Metabolism Disorders; Acid-Base Balance Disorder
Keywords: phosphorus; hemodialysis; bicarbonate; acidosis; alkalosis
MeSH Terms: conditions — Phosphorus Metabolism Disorders; Acidosis; Alkalosis

STUDY DESIGN:
Intervention Model Description: Blood acid-base and uremic solute levels were measured in twenty chronic HD patients during 4-hour treatments with A) constant Dbic of 35 mmol/L; B) Dbic of 35 mmol/L for the first two hours and 30 mmol/L for the second two hours; and C) Dbic of 30 mmol/L for the first 2 hours and 35 mmol/L later. Treatment interventions were fixed during a given week, arterial blood samples were obtained predialysis and every hour during the treatment, during the second and third treatments of the week.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: B) Dbic 35 -30 mmol/L C) Dbic 30- 35 mmol/L (Active Comparator): Week 1 - a constant Dbic 35 mmol/L -Treatment A. Week 2 - Dbic 35 mmol/L for the first two hours followed by 30 mmol/L for the remainder of the treatment- Treatment B.
  Week 3 - a constant Dbic 35 mmol/L (wash-out period). Week 4 - Dbic 30 mmol/L for the first two hours followed by 35 mmol/L for the remainder of the treatment -Treatment C.
  Interventions: Other: Group 1: B) Dbic 35 -30 mmol/L C) Dbic 30- 35 mmol/L
- Group 2: C) Dbic 30- 35 mmol/L B) Dbic 35 -30 mmol/L (Active Comparator): Week 1 - a constant Dbic 35 mmol/L -Treatment A. Week 2 - Dbic 30 mmol/L for the first two hours followed by 35 mmol/L for the remainder of the treatment- Treatment C.
  Week 3 - a constant Dbic 35 mmol/L (wash-out period). Week 4 - Dbic 35 mmol/L for the first two hours followed by 30 mmol/L for the remainder of the treatment -Treatment B.
  Interventions: Other: Group 2: C) Dbic 30 -35 mmol/L B) Dbic 35- 30 mmol/L

INTERVENTIONS:
Other: Group 1: B) Dbic 35 -30 mmol/L C) Dbic 30- 35 mmol/L — A change Dbic in a middle of hemodialysis
  Arms: Group 1: B) Dbic 35 -30 mmol/L C) Dbic 30- 35 mmol/L
Other: Group 2: C) Dbic 30 -35 mmol/L B) Dbic 35- 30 mmol/L — A change Dbic in a middle of hemodialysis
  Arms: Group 2: C) Dbic 30- 35 mmol/L B) Dbic 35 -30 mmol/L

SUMMARY:
Hyperphosphatemia is still an unresolved problem among hemodialysis patients and significantly increases the risk of death from cardiovascular diseases. Research to date has not answered the question of whether dialysate bicarbonate concentration profiling can improve phosphate removal and its concentration without negative impact on the acid-base balance. This study addressed this issue.

Twenty stable hemodialysis patients will enroll to a four-week study during which different dialysate bicarbonate concentration profiles will be used each week. Each patient will undergo the following profiles (one-week periods): Treatment A - stable dialysate bicarbonate concentration Dbic 35 mmol/L during the whole HD session, Treatment B - Dbic 35 mmol/L for the first two hours and Dbic 30 mmol/L for the next two hours and Treatment C - the opposite mid-HD change Dbic from 30 to 35 mmol/L and one week wash-out period between Treatment B and C. We will collect blood samples each hour during the session and one hour after HD completion.

ELIGIBILITY:
Inclusion Criteria:

* stable general condition
* hemodialysis more than 3 months
* Dialysis 3 times a week/ 4 hours +/- 20 minutes
* Dialysis with arterio-venous fistulas
* bicarbonate titer before hemodialysis 22-24 mmol/l

Exclusion Criteria:

* diabetes mellitus
* cachexia
* inflamation processes
* usage of sevelamer last month
* utrafiltration during dialysis more than 2500 ml

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
The blood phosphorus concentration change in hemodialysis patient | 4 weeks
  The blood phosphorus concentration change in hemodialysis patient using dialysate bicarbonate profiling

SECONDARY OUTCOMES:
The maintaining the acid-base balance in accordance with applicable recommendations. | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Wieliczko Monika, Warsaw, Poland